CLINICAL TRIAL: NCT02743728
Title: Perinatal Stroke: Understanding Brain Reorganization Through Infant Neuroimaging and Neuromodulation
Brief Title: Perinatal Stroke: Understanding Brain Reorganization
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: Cerebral Palsy Alliance (Other); American Academy of Cerebral Palsy and Developmental Medicine (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: PT-2015-23643
Record Dates: First submitted 2016-02-19; First posted 2016-04-19 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Stroke; Hemiparesis
Keywords: perinatal stroke; transcranial magnetic stimulation; magnetic resonance imaging; diffusion tensor imaging; non-invasive brain stimulation; infant
MeSH Terms: conditions — Stroke; Paresis | interventions — Magnetic Resonance Imaging; Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Infants: Each infant will receive an Magnetic Resonance Imaging, then Transcranial Magnetic Stimulation Cortical Excitability testing, and General Movement Assessment. These 3 different components of the one arm in which all infants are involved will be collectively assessed.
  Interventions: Device: Magnetic Resonance Imaging; Device: Transcranial Magnetic Stimulation; Behavioral: General Movement Assessment

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Anatomical and Diffusion Tensor Imaging Analysis.
Device: Transcranial Magnetic Stimulation — Assessment of brain (cortical) excitability
Behavioral: General Movement Assessment — Spontaneous movement assessment of infant while lying in unperturbed state.

SUMMARY:
The incidence of perinatal stroke is relatively common, as high as 1 in 2,300 births, but little is known about the resulting changes in the brain that eventually manifest as cerebral palsy (CP). Motor signs that indicate the infant is beginning to develop CP often do not become evident for several months after the diagnosis of perinatal stroke which delays therapy. The main purpose of this study is to examine early brain reorganization in infants 3-12 months of age corrected for prematurity with perinatal stroke using magnetic resonance imaging (MRI) and non-invasive transcranial magnetic stimulation (TMS). In addition, the association between the brain reorganization and motor outcomes of these infant participants will be identified.

In this study, the MRI scans will include diffusion tensor imaging (DTI) - an established method used to investigate the integrity of pathways in the brain that control limb movement. Infants will be scanned during nature sleeping after feeding. The real scanning time will be less than 38 minutes. TMS is a painless, non-surgical brain stimulation device which uses principles of electromagnetic induction to excite cortical tissue from outside the skull. Using TMS as a device to modulate and examine cortical excitability in children with hemiparetic CP and in adults has been conducted previously.

In this infant study, we will assess cortical excitability from the motor cortex of both the ipsilesional and contralesional hemispheres under the guidance of a frameless stereotactic neuronavigation system. Additionally, the investigators will assess infants' movement quality using an age-appropriate standardized movement assessment. This will allow the investigators to examine the relationship between measures of motor pathway integrity and early signs of potential motor impairment. We will longitudinally follow enrolled infants, and complete repeat assessments at 12- and 24-months corrected age to assess how infants develop over time after perinatal stroke. The remote follow-up will occur at 5 years or less.

DETAILED DESCRIPTION:
Understanding the early brain reorganization before the brain has not yet largely reorganized is critical for developing efficacious early intervention. As a unique aspect of investigation, this study will combine Magnetic Resonance Imaging (MRI)/ Diffusion Tensor Imaging (DTI) and TMS to provide an additional opportunity to assess both the cortical excitability and corticospinal tract (CST) integrity in infants with perinatal stroke.

Identifying the association between laboratory assessment results and developmental outcomes is also critical. This study is to use MRI/DTI and TMS to comprehensively examine both the CST integrity and cortical excitability in infants following perinatal stroke, and to identify association with motor outcome as evaluated by movement assessment.

ELIGIBILITY:
Inclusion Criteria for Pilot Study:

* Birth diagnosis of unilateral perinatal stroke by cranial ultrasound, computer tomography (CT) or magnetic resonance imaging (MRI)
* Corrected gestational age between 3 and 24 months of age for both infants with stroke and typically developing infants

Exclusion Criteria for Pilot Study :

* Metabolic Disorders
* Neoplasm
* Disorders of Cellular Migration and Proliferation
* Acquired Traumatic Brain Injury
* Received surgeries that may constraint current spontaneous movements
* Indwelling metal or incompatible medical devices
* Received surgeries that may constraint current spontaneous movements
* Other neurologic disorders unrelated to stroke
* Small for gestational age (SGA): Infants are smaller in size than normal for the gestational age
* Apneic episodes and syncope (known heart defects) for the safety of participants in the stud.
* Genetic disorders
* Uncontrolled seizures

Additional Inclusion Criteria for Follow-up Study:

- Previous participation in pilot study

Additional Exclusion Criteria for Follow-up Study:

- Lack of wireless internet access or computer to participate in virtual Zoom call

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The pilot study portion will recruit infants with unilateral perinatal stroke between 3 to 5 months of corrected age to understand their brain reorganization after stroke.
  The follow-up study portion will recruit children aged 5 years or younger who have been diagnosed with perinatal stroke and who participated in the pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette T Gillick, PhD, MSPT, PT, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Lehman LL, Rivkin MJ. Perinatal arterial ischemic stroke: presentation, risk factors, evaluation, and outcome. Pediatr Neurol. 2014 Dec;51(6):760-8. doi: 10.1016/j.pediatrneurol.2014.07.031. Epub 2014 Aug 14. PMID 25444092
- [Background] Eyre JA, Taylor JP, Villagra F, Smith M, Miller S. Evidence of activity-dependent withdrawal of corticospinal projections during human development. Neurology. 2001 Nov 13;57(9):1543-54. doi: 10.1212/wnl.57.9.1543. PMID 11706088
- [Background] Chen CY, Tafone S, Lo W, Heathcock JC. Perinatal stroke causes abnormal trajectory and laterality in reaching during early infancy. Res Dev Disabil. 2015 Mar;38:301-8. doi: 10.1016/j.ridd.2014.11.014. Epub 2015 Jan 9. PMID 25577180
- [Background] Thelen E, Corbetta D, Spencer JP. Development of reaching during the first year: role of movement speed. J Exp Psychol Hum Percept Perform. 1996 Oct;22(5):1059-76. doi: 10.1037//0096-1523.22.5.1059. PMID 8865616
- [Background] Einspieler C, Prechtl HF. Prechtl's assessment of general movements: a diagnostic tool for the functional assessment of the young nervous system. Ment Retard Dev Disabil Res Rev. 2005;11(1):61-7. doi: 10.1002/mrdd.20051. PMID 15856440
- [Background] Eyre JA, Miller S, Clowry GJ, Conway EA, Watts C. Functional corticospinal projections are established prenatally in the human foetus permitting involvement in the development of spinal motor centres. Brain. 2000 Jan;123 ( Pt 1):51-64. doi: 10.1093/brain/123.1.51. PMID 10611120
- [Background] Eyre JA, Smith M, Dabydeen L, Clowry GJ, Petacchi E, Battini R, Guzzetta A, Cioni G. Is hemiplegic cerebral palsy equivalent to amblyopia of the corticospinal system? Ann Neurol. 2007 Nov;62(5):493-503. doi: 10.1002/ana.21108. PMID 17444535
- [Background] Gillick BT, Krach LE, Feyma T, Rich TL, Moberg K, Menk J, Cassidy J, Kimberley T, Carey JR. Safety of primed repetitive transcranial magnetic stimulation and modified constraint-induced movement therapy in a randomized controlled trial in pediatric hemiparesis. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S104-13. doi: 10.1016/j.apmr.2014.09.012. Epub 2014 Oct 2. PMID 25283350
- [Background] Gillick BT, Krach LE, Feyma T, Rich TL, Moberg K, Thomas W, Cassidy JM, Menk J, Carey JR. Primed low-frequency repetitive transcranial magnetic stimulation and constraint-induced movement therapy in pediatric hemiparesis: a randomized controlled trial. Dev Med Child Neurol. 2014 Jan;56(1):44-52. doi: 10.1111/dmcn.12243. Epub 2013 Aug 21. PMID 23962321
- [Background] Kirton A, Chen R, Friefeld S, Gunraj C, Pontigon AM, Deveber G. Contralesional repetitive transcranial magnetic stimulation for chronic hemiparesis in subcortical paediatric stroke: a randomised trial. Lancet Neurol. 2008 Jun;7(6):507-13. doi: 10.1016/S1474-4422(08)70096-6. Epub 2008 May 1. PMID 18455961
- [Background] Narayana S, Rezaie R, McAfee SS, Choudhri AF, Babajani-Feremi A, Fulton S, Boop FA, Wheless JW, Papanicolaou AC. Assessing motor function in young children with transcranial magnetic stimulation. Pediatr Neurol. 2015 Jan;52(1):94-103. doi: 10.1016/j.pediatrneurol.2014.08.031. Epub 2014 Sep 18. PMID 25439485
- [Background] van de Ruit M, Perenboom MJ, Grey MJ. TMS brain mapping in less than two minutes. Brain Stimul. 2015 Mar-Apr;8(2):231-9. doi: 10.1016/j.brs.2014.10.020. Epub 2014 Nov 8. PMID 25556004
- [Derived] Kowalski JL, Hickey M, Rao R, Georgieff MK, Chen M, Gillick BT. Safety of single-pulse TMS in two infants with implanted patent ductus arteriosus closure devices. Brain Stimul. 2020 May-Jun;13(3):861-862. doi: 10.1016/j.brs.2020.03.007. Epub 2020 Mar 14. No abstract available. PMID 32289718

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Infants
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants are included in these analyses.
Arm/Group | All Infants
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Cortical Excitability MEP Amplitude (µV)
Description: Cortical excitability of ipsilesional and contralesional hemispheres assessed by transcranial magnetic stimulation (TMS) in infants with perinatal stroke.
  TMS will be used to assess cortical excitability through electromagnetic depolarization of targeted cortical neurons through painless pulses delivered over the scalp. The estimated time of TMS assessment is around 2 hours during Visit 2. Outcome is reported as MEP amplitude in units of microvolts (µV).
Time Frame: 2 hours
Population: Of the 20 enrolled infants, 11 infants participated in TMS. 3 of the 11 infants participated in TMS sessions at two different timepoints; therefore, 14 datasets for TMS outcome measures (MEP amplitude (Outcome 1), Resting Motor Threshold (Outcome 2) were analyzed.
Measure: Median (Full Range); unit: µV
Arm/Group | All Infants
Number analyzed (Participants) | 14
µV | 325 [50 to 500]

2. Primary Outcome: Cortical Excitability Percentage of Maximum
Description: Cortical excitability of ipsilesional and contralesional hemispheres assessed by transcranial magnetic stimulation (TMS) in infants with perinatal stroke.
  TMS will be used to assess cortical excitability through electromagnetic depolarization of targeted cortical neurons through painless pulses delivered over the scalp. The estimated time of TMS assessment is around 2 hours during Visit 2. The outcome of motor threshold will be reported as the percentage of maximum stimulator output.
Time Frame: 2 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: %MSO
Arm/Group | All Infants
Number analyzed (Participants) | 14
%MSO | 70 [50 to 95]

3. Secondary Outcome: General Movement Assessment
Description: Movement quality will be assessed by general movement assessment (GMA). GMA requires 5-10 minutes videotaping when infants are placed in spine position for scoring. Infants are scores categorically as typical (present fidgety movements) or atypical (absent, sporadic, or abnormal fidgety movements). Outcome is reported as the number of typical infants and number of atypical infants.
Time Frame: 15 minutes
Population: Of the 20 enrolled infants, 12 were able to complete the General Movements Assessment (GMA). The GMA was only completed if infants were between 3-5 months of age at the time of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | All Infants
Number analyzed (Participants) | 12
Participants
  Typical | 8
  Atypical | 4

4. Secondary Outcome: Adverse Events
Description: Recording of adverse events will take place during TMS cortical mapping and MRI scanning of infants with perinatal stroke. Assessment of vital signs changes and pain/stress responses during both MRI and TMS assessment during visit 1 and visit 2.
  Outcome is reported as the number of adverse events recorded.
Time Frame: 2 days
Population: Of the 20 enrolled infants, 13 infants participated in either MRI or TMS (during which adverse events were recorded).
Measure: Number; unit: # Adverse Events
Arm/Group | All Infants
Number analyzed (Participants) | 13
# Adverse Events | 0

5. Secondary Outcome: Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT)
Description: The PEDI-CAT uses Item Response Theory statistical models to estimate a child's ability from a minimal number of items. Three functional domains will be assessed. The PEDI-CAT software provides normative standard scores presented as T scores and age percentile ranges to assess daily activities, mobility, and social/cognitive function. Outcome is reported as the mean score generated by the PEDI-CAT software.
  Scores are based on t-test values and do not have a unit of measure or a defined range.
  Higher scores indicate greater deviation from the standardized mean score.
Time Frame: 15 minutes
Population: Of the 20 enrolled infants, 6 infants participated in remote follow-up and were assessed with the PEDI-CAT.
Measure: Mean (Full Range); unit: normative age percentiles
Arm/Group | All Infants
Number analyzed (Participants) | 6
normative age percentiles
  Daily Activities | 46 [1 to 87]
  Mobility | 42 [1 to 78]
  Social/Cognitive | 38 [2 to 62]

ADVERSE EVENTS:
Time Frame: Recording of adverse events will take place during TMS cortical mapping and MRI scanning of infants with perinatal stroke. Assessment of vital signs changes and pain/stress responses during both MRI and TMS assessment during visit 1 and visit 2.
Arm/Group | All Infants
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/28/NCT02743728/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT02743728/ICF_001.pdf